CLINICAL TRIAL: NCT01532791
Title: Mitochondrial Encephalomyopathies and Mental Retardation: Investigations of Clinical Syndromes Associated With MtDNA Point Mutations
Brief Title: Natural History Study - Mitochondrial Disease
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michio Hirano, MD, Professor of Neurology, Columbia University
Other Study IDs: AAAB1425; 5P01HD032062 (NIH)
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: MELAS or m.3243 A>G Mitochondrial DNA Mutation Carrier
Keywords: MELAS; mitochondrial DNA mutation; mtDNA mutation; mitochondrial DNA; mitochondria; m.3243A>G mutation
MeSH Terms: conditions — MELAS Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — skin fibroblast blood urine buccal cells hair samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mtDNA mutation: m.3243 A>G carriers and their maternal relatives Other mutations in the mitochondrial genome may be included
- Control: controls (people not maternally related to mutation carriers) Preference is for married in relatives

SUMMARY:
Carriers of the m.3242A>G mutation often have clinical symptoms which can include migraines, seizures, strokes, hearing loss, balance issues, gastrointestinal issues, and many other symptoms. The investigators would like to learn more about these disorders and have designed a "Natural History Study" to monitor these conditions over time so that physicians and scientists can not only understand the problems that patients have, but work on developing treatments. The focus of the current work is to evaluate known mutation carriers of the m.3243A>G (mitochondrial DNA) and their maternal relatives (carrier status not a requirement for participation). Paternal relatives will serve as controls. This study involves no treatment.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the neurological and biochemical consequences of the m.3243 A>G mutation. Mitochondria are the powerhouses of the cell and are controlled by nuclear genetic material (DNA) and mitochondrial (mt) DNA. Mitochondrial DNA mutations impair mitochondrial function, and cause cellular energy failure. These mutations, when present in high abundance, cause neurological signs and symptoms that are clinically obvious. The investigators hypothesize that these mutations, when present in lesser abundance, will cause measurable alterations in the patient's neuropsychological profile and cerebral energy profile. This study does not involve any experimental or approved therapy. The investigators will evaluate the patient's condition with blood/urine tests, neurological exam, MRI/MRS, questionnaires, motor skills functioning, serum and urine biomarkers, and genetic testing.

ELIGIBILITY:
Inclusion Criteria:

Known carrier of a the m.3243 A>G mitochondrial mutation, ,or Maternally related to someone who carries the m.3243A>G mitochondrial mutation.

A family member who is not maternally related to someone who carries the m.3243A>G mitochondrial mutation

Exclusion Criteria:

* Younger than 4 years of age
* No confirmed m.3243 A>G mitochondrial DNA mutation in the family.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Carriers of the m.3243A>G mitochondrial DNA point mutation, and their maternal relatives (carrier status documentation not required.). All patients suspected of having an mtDNA point mutation regardless of age, health status, gender, race, or ethnicity will be evaluated. The minimal age of entry into the study will be 4 years or older. We will also evaluate controls (often these are married in relatives).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2004-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
MRI/MRS | 2-3 years
  Evaluate structure and function in brain and muscle

SECONDARY OUTCOMES:
Biomarkers | 2-3 years
  Evaluate various biomarkers of disease progression
Motor skills | 2-3 years
  6 minute walk test to evaluate motor skills
Cognitive function | 2-3 years
  Evaluate cognitive function through neuropsychological testing
Clinical symptoms | 2-3 years
  Evaluate clinical symptoms through medical history questionnaires and physical exam
Mutation load | 2-3 years
  Evaluate heteroplasmy through blood,urine and skin fibroblast evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Principal Investigator — mh29@cumc.columbia.edu
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
When applicable, manuscript(s) regarding data will be submitted for publication

REFERENCES:
- [Background] Weiduschat N, Kaufmann P, Mao X, Engelstad KM, Hinton V, DiMauro S, De Vivo D, Shungu D. Cerebral metabolic abnormalities in A3243G mitochondrial DNA mutation carriers. Neurology. 2014 Mar 4;82(9):798-805. doi: 10.1212/WNL.0000000000000169. Epub 2014 Jan 29. PMID 24477106
- [Background] Kaufmann P, Engelstad K, Wei Y, Kulikova R, Oskoui M, Sproule DM, Battista V, Koenigsberger DY, Pascual JM, Shanske S, Sano M, Mao X, Hirano M, Shungu DC, Dimauro S, De Vivo DC. Natural history of MELAS associated with mitochondrial DNA m.3243A>G genotype. Neurology. 2011 Nov 29;77(22):1965-71. doi: 10.1212/WNL.0b013e31823a0c7f. Epub 2011 Nov 16. PMID 22094475
- [Background] Mehrazin M, Shanske S, Kaufmann P, Wei Y, Coku J, Engelstad K, Naini A, De Vivo DC, DiMauro S. Longitudinal changes of mtDNA A3243G mutation load and level of functioning in MELAS. Am J Med Genet A. 2009 Feb 15;149A(4):584-7. doi: 10.1002/ajmg.a.32703. PMID 19253345
- [Background] Kaufmann P, Engelstad K, Wei Y, Kulikova R, Oskoui M, Battista V, Koenigsberger DY, Pascual JM, Sano M, Hirano M, DiMauro S, Shungu DC, Mao X, De Vivo DC. Protean phenotypic features of the A3243G mitochondrial DNA mutation. Arch Neurol. 2009 Jan;66(1):85-91. doi: 10.1001/archneurol.2008.526. PMID 19139304
- See also: general website for our available clinical studies — http://www.giblinlab.org